CLINICAL TRIAL: NCT06576804
Title: Effects of Concentric and Eccentric Exercise Regimens on Bioenergetic Efficiency of Lymphocytes in Sedentary Males
Brief Title: Eccentric Cycling Exercise on Mitochondrial Function of Lymphocyte
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202100004A3
Record Dates: First submitted 2024-08-20; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Eccentric Exercise Training
Keywords: Eccentric cycling; Mitochondria; Lymphocyte

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eccentric cycling training (Experimental): Moderate to high intensity cycling training in eccentric type
  Interventions: Behavioral: Eccentric cycling training
- Concentric cycling training (Experimental): Moderate to high intensity cycling training in concentric type (intensity matched the eccentric training)
  Interventions: Behavioral: Concentric cycling training
- Control group (No Intervention): without receiving any exercise training

INTERVENTIONS:
Behavioral: Eccentric cycling training — Performed exercise training 5 days a week for 6 weeks on an eccentric ergometer.
  Each training session: 5 min at 30% of maximal workload (Wmax) for warmed up and cold down and 30 min the main training phase.
  Intensity: Firstly, set at 60% Wmax, and progressively increased 5% per week
  Arms: Eccentric cycling training
Behavioral: Concentric cycling training — Performed exercise training 5 days a week for 6 weeks on an eccentric ergometer.
  Each training session: 5 min at 30% of maximal workload (Wmax) for warmed up and cold down and 30 min the main training phase.
  Intensity: Firstly, set at 60% Wmax, and progressively increased 5% per week
  Arms: Concentric cycling training

SUMMARY:
Eccentric cycling exercise (ECE) features lower metabolic demand and higher improvement of muscle strength compared to traditional concentric cycling exercise (CCE). Mitochondria can regulate energy metabolism and adaptive immune quality in T lymphocytes. However, the effects of ECE on mitochondrial functions in T-lymphocytes have not yet been established.

Method: A total of 33 healthy sedentary males were randomized and divided into ECE (n=11), CCE (n=11), and control groups (n=11). These subjects progressively performed CCE or ECE from 60% to 80% maximal workload on a bicycle ergometer for 40 min/day, 5 days/week for 6 weeks. A graded exercise testing and an isokinetic strength test were conducted to evaluate cardiopulmonary fitness and muscle strength, respectively. Phenotypes and mitochondrial respiratory capacity in T lymphocyte were analyzed using flow cytometry and high-resolution respirometer, respectively.

DETAILED DESCRIPTION:
Eccentric exercise training (EET) increases physical performance while having lower metabolic demand than concentric exercise training (CET).

Mitochondria of lymphocytes are essential for cell proliferation, death, and differentiation, and play a critical role in establishing lymphocyte phenotypes and their functions.

Whether EET influences lymphocyte bioenergetic efficiency remains unclear. The study was to investigate the effects of ECE and CCE regimens on adaptive immune functions and mitochondrial bioenergetics of T lymphocytes in sedentary males.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary lifestyle.
2. Nonsmokers, nonusers of medications/vitamins.
3. No any cardiopulmonary/hematological risks.

Exclusion Criteria:

1. Have regular exercise habits (i.e., exercise frequency once per week, duration >20 min).
2. Have retabolic or musculoskeletal disease.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Mitochondrial function of lymphocyte | 12 weeks
  Evaluate bioenergetic health index (BHI) of mitochondria in lymphocyte by using a high resolution respirometer.

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 12 weeks
  The graded exercise test (GXT) on a bicycle ergometer was performed. The GXT comprised 2 min of unloaded pedaling followed by a continuous increase in the work rate of 30 watt per 3-minute until exhaustion (i.e., progressive exercise to maximal O2 consumption)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] LaStayo PC, Ewy GA, Pierotti DD, Johns RK, Lindstedt S. The positive effects of negative work: increased muscle strength and decreased fall risk in a frail elderly population. J Gerontol A Biol Sci Med Sci. 2003 May;58(5):M419-24. doi: 10.1093/gerona/58.5.m419. PMID 12730250
- [Result] Hody S, Croisier JL, Bury T, Rogister B, Leprince P. Eccentric Muscle Contractions: Risks and Benefits. Front Physiol. 2019 May 3;10:536. doi: 10.3389/fphys.2019.00536. eCollection 2019. PMID 31130877
- [Result] Touron J, Costes F, Coudeyre E, Perrault H, Richard R. Aerobic Metabolic Adaptations in Endurance Eccentric Exercise and Training: From Whole Body to Mitochondria. Front Physiol. 2021 Jan 27;11:596351. doi: 10.3389/fphys.2020.596351. eCollection 2020. PMID 33584331
- [Result] Tsai HH, Chang SC, Chou CH, Weng TP, Hsu CC, Wang JS. Exercise Training Alleviates Hypoxia-induced Mitochondrial Dysfunction in the Lymphocytes of Sedentary Males. Sci Rep. 2016 Oct 12;6:35170. doi: 10.1038/srep35170. PMID 27731374